CLINICAL TRIAL: NCT01191853
Title: Cellular and Molecular Characterization of the Immune Response in Healthy NIH Employees at Baseline, and After Immunization With the H1N1 or Seasonal Influenza Vaccines
Brief Title: Cellular and Molecular Characterization of the Immune Response in Healthy NIH Employees atBaseline, and After Immunization With the H1N1 or Seasonal Influenza Vaccines
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090239; 09-H-0239
Record Dates: First submitted 2010-08-28; First posted 2010-08-31 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-12-15

CONDITIONS: Healthy Volunteers; Influenza
Keywords: Post Swine Flu Blood Samples; Biologic Sample Collection; Laboratory Research Samples; Natural History; Healthy Volunteer; HV
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy volunteers: Healthy volunteers will have blood drawn before and after seasonal flu vaccination

SUMMARY:
Background:

- Seasonal influenza is a major health problem whose impact is typically reduced by vaccination. The H1N1 (swine flu) influenza virus is an emerging pathogen that has the potential to cause devastating illness and even death in the coming months. Currently, there are limited data on the cellular and molecular immune responses in adult recipients of either the seasonal or the H1N1 influenza vaccines.

Objectives:

- To obtain blood and nasal wash samples and perform laboratory studies to characterize the immune response in healthy adult volunteers at baseline and after immunization with the seasonal or H1N1 influenza vaccines.

Eligibility:

- Adult employees at least 18 years of age of the NIH Clinical Center who are deemed healthy by a brief medical history and physical examination and routine blood testing.

Design:

* Before the start of the influenza season, volunteers will receive either the seasonal influenza vaccine or the H1N1 vaccine when it becomes available. If the H1N1 vaccine is available at the start of the season, volunteers will receive both the seasonal vaccine and the H1N1 vaccine.
* Blood will be drawn over an 8-week period. Volunteers must not eat anything for 8 hours prior to the blood draw. The sequence of the blood draws is as follows: 2 weeks before vaccination; right before vaccination; and 1, 7, 14, 28, and 60 days after vaccination.
* Two to four nasal washings will be collected by a nurse before volunteers receive the vaccination(s) and 28 days after the vaccination.
* Prevaccine and postvaccine blood and nasal wash samples will be compared to determine volunteers immune responses.
* Research samples will be stored indefinitely and will be used strictly for laboratory experiments.

DETAILED DESCRIPTION:
Seasonal influenza is a major health problem whose impact is typically reduced by vaccination. The H1N1 (swine flu) influenza virus is an emerging pathogen which has the potential to cause devastating morbidity and mortality in the coming months. In June 2009, the World Health Organization declared the H1N1 outbreak to be a global pandemic. At present there are limited data on the cellular and molecular immune responses in adult recipients of either the seasonal or the H1N1 influenza vaccines.

Therefore, the Center for Human Immunology, Autoimmunity, and Inflammatory Diseases proposes this protocol designed to obtain blood from healthy adult subjects (NIH employees) prior to vaccination and then at various time points after receiving the FDA-licensed seasonal and H1N1 influenza vaccine. These samples will be used to perform a comprehensive and detailed analysis of the immune system at baseline and in response to vaccination. To our knowledge, this protocol will be the first study to characterize the human cellular and molecular immune system parameters, or immunome, in a large number of healthy adults (NIH employees). This information may be useful in designing newer, more effective vaccines to prevent the spread of H1N1 influenza.

The primary objective is to perform laboratory studies to characterize the immune response in healthy adult volunteers at baseline and after immunization with the seasonal or H1N1 influenza vaccines. Primary endpoint is the results of the research laboratory assessments. As samples will be stored indefinitely, the time frame for primary endpoint is indefinite.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. NIH employees scheduled to receive the Influenza and H1N1 vaccines through OMS.
  2. Health status confirmed by History, Physical Exam and blood work through the CHI Screening Protocol.
  3. Age 18 years and older (no upper limit).
  4. Able to comprehend the investigational nature of the protocol and provide informed consent.

EXCLUSION CRITERIA:

1. Recipient of another vaccine or immune modulating drug within 6 months prior to study entry.
2. Severe allergies to eggs or their products.
3. Prior severe reactions to vaccines.
4. Participation on any blood collection or blood donation procedure during study participation.
5. Current pregnancy (women of child bearing potential must have a negative serum pregnancy test done on screening within 1 week of protocol accrual).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy NIH Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2009-09-18

PRIMARY OUTCOMES:
Analysis of immune response after vaccine | continuous
  Immune response to vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Pamela L Schwartzberg, Ph.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Thompson WW, Shay DK, Weintraub E, Brammer L, Cox N, Anderson LJ, Fukuda K. Mortality associated with influenza and respiratory syncytial virus in the United States. JAMA. 2003 Jan 8;289(2):179-86. doi: 10.1001/jama.289.2.179. PMID 12517228
- [Background] Zimmer SM, Burke DS. Historical perspective--Emergence of influenza A (H1N1) viruses. N Engl J Med. 2009 Jul 16;361(3):279-85. doi: 10.1056/NEJMra0904322. Epub 2009 Jun 29. No abstract available. PMID 19564632
- [Background] Taubenberger JK, Morens DM. 1918 Influenza: the mother of all pandemics. Emerg Infect Dis. 2006 Jan;12(1):15-22. doi: 10.3201/eid1201.050979. PMID 16494711
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-H-0239.html